CLINICAL TRIAL: NCT07398469
Title: A Longitudinal Online Survey of Patient-Reported Changes in Postpartum Depression Symptoms Following Zuranolone Use
Brief Title: A Long-Term Study of Patient-Reported Changes in Postpartum Depression Symptoms in People Starting Zuranolone
Status: Recruiting | Type: Observational
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Other Study IDs: US-ZRN-12376
Record Dates: First submitted 2026-02-04; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Postpartum Depression
MeSH Terms: conditions — Depression, Postpartum | interventions — zuranolone

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Zuranolone: Participants who are prescribed zuranolone for PPD will be contacted for enrolment.
  Interventions: Drug: Zuranolone

INTERVENTIONS:
Drug: Zuranolone — Administered orally
  Other Names: Zurzuvae; BIIB125

SUMMARY:
In this study, researchers will learn how postpartum depression symptoms may change after people first start taking zuranolone. This is a drug available for doctors to prescribe for people with postpartum depression, also known as PPD. After giving birth, people with PPD can suffer from symptoms like tiredness, sadness, and a loss of interest in their daily activities.

This is known as an "observational" study, which collects health information about study participants without changing their medical care. Participants for this study will be found in the United States using a database from Accredo Specialty Pharmacy. This will include anyone who has a new prescription for zuranolone and were pregnant in the last 12 months before joining the study.

The main goal of this study is to learn more about how zuranolone affects the participants' PPD symptoms. This will be done using a questionnaire called the Edinburgh Postnatal Depression Scale, also known as the EPDS.

The main question that researchers want to answer is:

• Do PPD symptoms change after treatment with zuranolone based on EPDS scores measured at Day 15?

Researchers will also learn about :

* Changes in participants' EPDS scores at Day 45 and Day 90 in the study
* Changes in EPDS scores at Day 15, Day 45, and Day 90 in a group of participants who have moderately severe PPD before starting zuranolone
* How many participants breastfeed their babies while taking zuranolone
* How many participants report not starting new medicine after finishing their zuranolone treatment

The study will be done as follows:

* People with PPD who get a new zuranolone prescription through Accredo Specialty Pharmacy will be contacted by email or phone to ask them about their interest in participating in the study.
* Before taking their first dose of zuranolone, participants will be asked to answer written questions about their symptoms using the online EPDS survey. They will also answer other survey questions about their background, environment, and general health information. Participants must take their first dose of zuranolone within 7 days of joining the study.
* Participants will then be asked to answer questions using the EPDS survey, 15 days, 45 days, and 90 days after taking the first dose of zuranolone. Each survey will take about 10-15 minutes to finish.

DETAILED DESCRIPTION:
The primary objective of this study is to assess the reduction in Postpartum Depression (PPD) symptoms via the Edinburgh Postnatal Depression Scale (EPDS) at Day 15 in study participants. The secondary objectives are to assess the reduction in PPD symptoms via the EPDS at Day 45 and Day 90 in study participants, reduction in PPD symptoms via the EPDS at Day 15,Day 45, and Day 90 in a subgroup of participants with moderate PPD at baseline, to assess breastfeeding status during treatment with zuranolone as reported at Day 45 and to characterize treatment usage across the 90-day period via self-reported survey questions.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants with a prescription for zuranolone via Accredo Specialty Pharmacy.
* Recent pregnancy in the last 12 months.
* Confirmed diagnosis of PPD.
* Able to complete the questionnaires by themselves in English.

Key Exclusion Criteria:

* Prior fill of zuranolone or brexanolone in last 12 months.
* Participants who have taken 1 or more doses of zuranolone at the time of study screening.
* Current or history of bipolar disorder.
* Failure to complete baseline (Day 0) surveys.
* Declined to consent.
* Pregnancy that ended more than 12 months ago.

Note: Other protocol-defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Participants prescribed zuranolone who consent to participate in this study and meet all of the inclusion criteria, none of the exclusion criteria, and complete baseline (Day 0) will be considered enrolled in this study.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-12-22 (Actual); Primary Completion 2027-03-29 (Estimated); Study Completion 2027-03-29 (Estimated)

PRIMARY OUTCOMES:
Change From Baseline in the Edinburgh Postnatal Depression Scale (EPDS) Score at Day 15 | Baseline (Day 0), Day 15
  EPDS is a 10-item self-report questionnaire used for the assessment of PPD symptoms. Each item is scored from 0-3, with a total score range of 0-30. Higher scores indicate more severe depressive symptoms.

SECONDARY OUTCOMES:
Change From Baseline in the EPDS Score at Days 45 and 90 | Baseline (Day 0), Days 45 and 90
  EPDS is a 10-item self-report questionnaire used for the assessment of PPD symptoms. Each item is scored from 0-3, with a total score range of 0-30. Higher scores indicate more severe depressive symptoms.
Change From Baseline in the EPDS Score at Days 15, 45, and 90 in Participants With Moderate Severity | Baseline (Day 0), Days 15, 45 and 90
  EPDS is a 10-item self-report questionnaire used for the assessment of PPD symptoms. Each item is scored from 0-3, with a total score range of 0-30. Higher scores indicate more severe depressive symptoms.
Number of Participants With no New Initiation of Medication After Completion of Zuranolone | At Days 45 and 90
  This outcome measure will be self-reported by participants.
Number of Participants With Moderate Postpartum Depression (PPD) Severity and no New Initiation of Medication After Completion of Zuranolone | At Days 45 and 90
  This outcome measure will be self-reported by participants.
Number of Participants Feeding Their Baby Breastmilk as Usual While Taking Zuranolone | At Day 45
  This outcome measure will be self-reported by participants.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Biogen, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on htps://www.biogentrialtransparency.com/
URL: https://vivli.org/